CLINICAL TRIAL: NCT07226921
Title: Language Control Across Comprehension and Production in Unimodal and Bimodal Bilinguals
Brief Title: Language Control Across Modalities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Chuchu Li, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 806634; R01HD116841 (NIH)
Record Dates: First submitted 2025-11-06; First posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: language control; bilingual adults; reaction time

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Predictable one-language production & both-language comprehension (Experimental)
  Interventions: Behavioral: Predictability; Behavioral: language context
- Predictable both-language production & both-language comprehension (Experimental)
  Interventions: Behavioral: Predictability; Behavioral: language context
- Unpredictable one-language production & both-language comprehension (Experimental)
  Interventions: Behavioral: Predictability; Behavioral: language context
- Single language comprehension and production (No Intervention)

INTERVENTIONS:
Behavioral: Predictability — Whether the task of the next trial (comprehension or production) is predictable
  Arms: Predictable both-language production & both-language comprehension; Predictable one-language production & both-language comprehension; Unpredictable one-language production & both-language comprehension
Behavioral: language context — whether both languages or only one language is involved in the current block
  Arms: Predictable both-language production & both-language comprehension; Predictable one-language production & both-language comprehension; Unpredictable one-language production & both-language comprehension

SUMMARY:
This study aims to investigate how unimodal bilinguals who speak two languages and bimodal bilinguals who speak one language and sign another control languages across comprehension and production. Participants will complete different language tasks (e.g., classify a word, name a picture) in different languages, and their behavioral performance will be assessed, including accuracy and reaction time.

ELIGIBILITY:
Inclusion Criteria:

* Proficient in both Mandarin and English, or proficiency in both ASL and English

Exclusion Criteria:

* Know a third language better than Mandarin/English or better than ASL/English
* With language disorder or other neurological disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2030-05-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Switch costs in different contexts | An average of one year for each condition

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD, San Diego, California, United States